CLINICAL TRIAL: NCT06874686
Title: Minimally Invasive Laparoscopic Surgery for Hirschsprung's Disease: a Retrospective Study on Patient Safety Profiles, Effectiveness, and Short-term Functional Outcomes
Brief Title: Minimally Invasive Surgical Intervention for Hirschsprung's Disease in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Nguyen Thanh Quang, Principle Investigator, National Children's Hospital, Vietnam
Other Study IDs: 1451_06/BVNTW-VNCSKTE
Record Dates: First submitted 2025-03-02; First posted 2025-03-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Hirschsprung Disease
Keywords: Aganglionic; Minimally invasive; Laparoscopic; Pediatric; Single incision; Hirschsprung; Hirschsprung disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MIS-Treated Hirschsprung Patients (2017-2023): Pediatric patients diagnosed with Hirschsprung's Disease, admitted to the National Children's Hospital between January 2017 and December 2023, exhibiting clinical signs and symptoms consistent with Hirschsprung disease, with imaging findings confirming the diagnosis.
  Interventions: Procedure: Minimally invasive laparoscopic pull-through surgery

INTERVENTIONS:
Procedure: Minimally invasive laparoscopic pull-through surgery — Pediatric patients diagnosed with Hirschsprung's Disease from 2017-2023 at the National Children's Hospital underwent two minimally invasive procedures: conventional laparoscopic pull-through (CLP) and single-incision laparoscopic pull-through (SILPS).
  CLP involves three to five small incisions for trocars, allowing laparoscopic visualization and instrument access. Pneumoperitoneum is established, and the aganglionic colon segment is identified and mobilized using laparoscopic energy devices. The rectum is dissected circumferentially to preserve mesenteric blood supply, and a transanal approach is used to excise the diseased segment, followed by coloanal anastomosis with absorbable sutures.
  SILPS follows the same principles but is performed through a single umbilical incision using a multi-port device for all instruments. This technique offers benefits like reduced scarring and less postoperative pain but requires advanced laparoscopic skills due to instrument crowding.

SUMMARY:
Hirschsprung's disease (HD) is a congenital disorder characterized by the absence of enteric ganglion cells in the distal bowel, leading to functional obstruction, delayed meconium passage in neonates, and chronic defecation difficulties. Surgical intervention is required to remove the aganglionic segment, with minimally invasive laparoscopic techniques increasingly preferred over open surgery due to reduced postoperative complications, shorter hospital stays, and faster recovery. Since 2012, the National Children's Hospital has pioneered the routine use of single-incision laparoscopic surgery (SILS) for HD in Vietnam. However, there is a lack of comprehensive analysis on the operative outcome in this large group of patients. This retrospective study aims to evaluate patient safety profiles, surgical effectiveness, and functional outcomes of minimally invasive laparoscopic procedures for HD performed at the National Children's Hospital between 2017 and 2023.

DETAILED DESCRIPTION:
Hirschsprung's disease (HD) is a congenital disorder caused by the absence of enteric ganglion cells in the distal bowel, leading to functional obstruction, delayed meconium passage in neonates, and defecation difficulties. If left untreated, HD can result in life-threatening complications such as Hirschsprung-associated enterocolitis and severe bowel dysfunction. Surgical intervention is necessary to remove the aganglionic segment and restore normal bowel function. In recent years, minimally invasive laparoscopic techniques have gained preference over open surgery due to their potential to reduce intraoperative blood loss, postoperative pain, surgical site infections, and overall hospital stay, while promoting faster recovery and improved cosmetic outcomes. The conventional 3 ports laparoscopic rectal pull-through technique has been widely used as the standard treatment for HD since its introduction in 1995. In 2010, the first case series of single-incision laparoscopic-assisted rectal pull-through (SILS) surgery for HD was reported. The study demonstrated that SILS is safe, yielding comparable surgical outcomes while reducing surgical trauma and enhancing cosmetic results.

Since 2012, the National Children's Hospital has been at the forefront of utilizing minimally invasive approaches for HD treatment in Vietnam, particularly through single-incision laparoscopic surgery (SILS) and conventional multi-port laparoscopic pull-through (CLP). However, despite the increasing adoption of these techniques, there remains a lack of comprehensive data on their surgical outcome, in a lower-middle-income country setting. Factors such as limited research funding, financial constraints preventing patients from accessing long-term follow-up care, and variability in postoperative management contribute to the gap in knowledge regarding these surgical approaches.

This retrospective study aims to systematically evaluate the safety profiles, clinical effectiveness, and short-term functional outcomes of minimally invasive laparoscopic procedures for HD performed at the National Children's Hospital between 2017 and 2023. Key parameters of analysis will include perioperative complications, length of hospital stay, surgical success rates, incidence of postoperative enterocolitis, fecal continence, bowel function recovery, and cost-effectiveness of the intervention. By providing a detailed assessment of these factors, this study seeks to optimize surgical management strategies, enhance postoperative care, and contribute to the growing body of evidence supporting minimally invasive surgical techniques for HD in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (under 18 years old) diagnosed with Hirschsprung's Disease, admitted to National Children's Hospital between January 2017 and December 2023.
* Patients exhibiting clinical signs and symptoms consistent with Hirschsprung's Disease, with imaging findings confirming the diagnosis. If imaging was inconclusive but clinical suspicion remained high, patients were still considered for surgical evaluation and management.
* Underwent minimally invasive laparoscopic pull-through surgery, either conventional multi-port (CLP) or single-incision (SILS).
* Postoperative Follow-up Data Availability: Patients with documented short-term postoperative outcomes, including bowel function recovery, complications, or reoperation rates.

Exclusion Criteria:

* Clinical instability requiring emergency open laparotomy due to peritonitis, intestinal perforation, or other life-threatening conditions.
* Biopsy findings inconsistent with Hirschsprung's Disease, ruling out the diagnosis.
* Incomplete Medical Records: Patients with missing key data, such as operative details, pathology reports, or follow-up outcomes, that could compromise study integrity

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study includes pediatric patients (<18 years) diagnosed with Hirschsprung's Disease, admitted to National Children's Hospital (2017-2023). Eligible patients exhibited clinical signs and symptoms, with imaging confirming the diagnosis or high clinical suspicion warranting surgery.
  All underwent minimally invasive laparoscopic pull-through surgery (CLP or SILS) with documented short-term postoperative outcomes.
  Exclusions include patients requiring emergency open laparotomy, those with biopsy findings inconsistent with Hirschsprung's Disease, or incomplete medical records.
  Data will be collected retrospectively to assess the safety and effectiveness of these surgical techniques.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2025-02 (Actual)

PRIMARY OUTCOMES:
Volume of Blood Loss | Perioperative
  The amount of blood lost during surgery will be measured in milliliters (mL) by collecting blood from suction devices, counting soaked surgical sponges, and assessing any other visible loss
Conversion to open surgery | Perioperative
  The proportion of cases in which single-incision laparoscopic surgery (SILS) could not be optimally completed and required conversion to open surgical techniques. Conversion may be necessitated by factors such as poor visualization, uncontrolled bleeding, adhesions, or patient-specific anatomical challenges. The outcome will be measured as the percentage of procedures requiring conversion during the perioperative period.
Operative time | Perioperative
  Total duration of the surgical procedure from skin incision to closure, measured in minutes.
Mortality and severe morbidity | Through study completion, an average of 5 years
  The incidence of mortality and severe postoperative complications following single-incision laparoscopic pull-through surgery. Severe morbidity includes life-threatening conditions such as sepsis, multi-organ failure, other major complications requiring intensive medical intervention, and death.
Early postoperative complications | Up to 8 weeks post-operation
  The incidence of early postoperative complications, including but not limited to bowel obstruction, surgical site infections, and Hirschsprung-associated enterocolitis (HAEC). Additional complications such as anastomotic leakage, prolonged ileus, or unexpected reoperation will also be monitored.
Time to return of bowel function | Up to 4 weeks post-operation
  The time from surgical intervention to the return of bowel function, defined as the first occurrence of spontaneous bowel movement or passage of flatus without the need for rectal stimulation or enemas
Rate of reoperation | Through study completion, an average of 5 years
  The proportion of patients who require an additional surgical intervention related to the initial procedure. This includes cases of anastomotic complications, bowel obstruction, stricture formation, or other postoperative issues necessitating reoperation.
Fecal Continence and Bowel Function Recovery | Through study completion, an average of 5 years
  Frequency of bowel movements, presence of soiling, need for enemas, and ability to maintain voluntary bowel control at follow-up visits.
Length of Hospital Stay | Up to 24 weeks post-operation
  The total number of days from admission to discharge after surgery, reflecting postoperative recovery and hospital resource utilization.

SECONDARY OUTCOMES:
Total cost of the Surgical Approach | Through study completion, an average of 5 years
  Total cost of hospitalization, medications, and additional treatments to assess the overall economic feasibility in a lower-middle-income setting.
Diagnostic predictive value of X-ray for Hirschsprung Disease | Perioperative
  This outcome measures the diagnostic accuracy of X-ray in detecting Hirschsprung disease by comparing its findings to biopsy results. It evaluates whether the resected bowel contains the aganglionic segment and assesses the completeness of aganglionic bowel resection. Diagnostic performance will be analyzed using sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Quang T Nguyen, M.D., Principal Investigator — Department of Pediatric Surgery, The National Hospital of Pediatrics, Hanoi, Vietnam
Locations (1):
- Department of Surgery, The National Children Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amiel J, Lyonnet S. Hirschsprung disease, associated syndromes, and genetics: a review. J Med Genet. 2001 Nov;38(11):729-39. doi: 10.1136/jmg.38.11.729. PMID 11694544
- [Background] Muensterer OJ, Chong A, Hansen EN, Georgeson KE. Single-incision laparoscopic endorectal pull-through (SILEP) for hirschsprung disease. J Gastrointest Surg. 2010 Dec;14(12):1950-4. doi: 10.1007/s11605-010-1299-3. Epub 2010 Aug 18. PMID 20717739
- [Background] Ure BM, Rintala RJ, Holschneider AM. Scoring postoperative results. Anorectal Malformations Child Embryol Diagnosis, Surg Treat Follow. 2006;351-9. . : . .
- [Background] Nguyen LT, Nguyen AT, Nguyen QT, Tran QA, Bui HD, Pham HD. Suspension sutures facilitate single-incision laparoscopic-assisted rectal pull-through for Hirschsprung disease. BMC Surg. 2021 May 31;21(1):274. doi: 10.1186/s12893-021-01260-w. PMID 34059040
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Xia X, Li N, Wei J, Zhang W, Yu D, Zhu T, Feng J. Single-incision laparoscopic versus conventional laparoscopic surgery for Hirschsprung's disease: A comparison of medium-term outcomes. J Pediatr Surg. 2016 Mar;51(3):440-3. doi: 10.1016/j.jpedsurg.2015.10.051. Epub 2015 Oct 24. PMID 26611332
- [Background] Zimmermann P, Martynov I, Perger L, Scholz S, Lacher M. 20 Years of Single-Incision-Pediatric-Endoscopic-Surgery: A Survey on Opinion and Experience Among International Pediatric Endosurgery Group Members. J Laparoendosc Adv Surg Tech A. 2021 Mar;31(3):348-354. doi: 10.1089/lap.2020.0797. Epub 2020 Dec 31. PMID 33395367
- [Background] Georgeson KE, Robertson DJ. Laparoscopic-assisted approaches for the definitive surgery for Hirschsprung's disease. Semin Pediatr Surg. 2004 Nov;13(4):256-62. doi: 10.1053/j.sempedsurg.2004.10.013. PMID 15660319
- [Background] Mayo Clinic. Hirschsprung's disease - Symptoms and causes 2021 . : . .
- [Background] Puri P, Nakamura H. Epidemiology and Clinical Characteristics of Hirschsprung's Disease. In: Hirschsprung's Disease and Allied Disorders . : . .
- [Background] LÊ NH. ĐÁNH GIÁ KẾT QUẢ PHẪU THUẬT BỆNH GIÃN ĐẠI TRỰC TRÀNG BẨM SINH Ở NGƯỜI LỚN TẠI BỆNH VIỆN VIỆT ĐỨC. 2020 . : . .
- [Background] Liu, M., Fang, Y., Zhang, B., Lin, Y., Li, O., Bai, J., … & Wu, D. (2020). Laparoscopic-assisted soave operation for the treatment of hirschsprung disease in children: 5 years of experience.. https://doi.org/10.21203/rs.3.rs-18886/v1 . : . .